CLINICAL TRIAL: NCT00152438
Title: Vasomotor Symptoms and Endothelial Function-A Randomized Placebo-controlled Trial of Oral Micronized Progesterone (Prometrium®)
Brief Title: Vasomotor Symptoms (VMS) Progesterone Study: Vasomotor Symptoms and Endothelial Function - Trial of Oral Micronized Progesterone
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C03-0088
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Menopause
Keywords: Vasomotor symptoms; Menopause
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral micronized progesterone
  Interventions: Drug: Oral Micronized Progesterone (Prometrium®)
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral Micronized Progesterone (Prometrium®) — 300 mg per day in 3 - 100 mg pills, to be taken in the evening immediately before sleep.
  Other Names: Oral micronized progesterone: Prometrium®, Uteroestan®
  Arms: 1
Other: Placebo — 3 identical placebo pills daily, no active ingredient.
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine the effects of a full dose (300 mg at hs) of oral micronized progesterone (OMP) on vasomotor symptoms [VMS] (hot flushes/night sweats), on forearm blood flow and on lipid levels and blood pressure in menopausal women without cardiovascular disease and with moderate to severe VMS.

The hypotheses are that progesterone will improve hot flushes, increase endothelium-dependent forearm blood flow and will decrease blood pressure without change in lipid levels.

DETAILED DESCRIPTION:
In this 4-month study, menopausal women are randomized to either placebo or oral micronized progesterone (Prometrium®). Participants maintain a daily diary to keep track of their vasomotor symptoms and other factors. Forearm blood flow will be assessed by venous occlusion plethysmography at baseline and after three months of therapy. Screening tests at baseline to rule out heart disease include measurement of blood pressure and heart rate, electrocardiogram (ECG) and blood tests - fasting blood glucose and lipid profile.

Collection of serum and plasma samples at baseline and end of therapy for analysis of cardiovascular markers (e.g., c-reactive protein) and clotting and fibrinolytic markers. Continued daily diary collection for one month after therapy discontinuation to look for possible rebound effects. Analysis of outcomes will be by analysis of covariates, with final value as the outcome, therapy as factor and baseline values as covariate.

ELIGIBILITY:
Inclusion Criteria:

1. Menopausal women (final menstrual period one or more but less than 10 years before)
2. No evidence of vascular disease (normal BP; without diabetes mellitus; normal cholesterol levels and non-smoker for at least a year; and normal ECG.)
3. Moderate to severe VMS during the day and night.

Exclusion Criteria:

1. Any menstruation in the preceding year.
2. History of hysterectomy without ovariectomy unless 60 years of age.
3. Use of ovarian hormone therapy (estrogen, progestin, progesterone or androgen) or selective estrogen receptor modulator (SERM) therapy (raloxifene or tamoxifen) in the preceding six months.
4. Body mass index (BMI) over 35 or less than 20.
5. Mean of several pre-treatment blood pressures over 145/95.
6. Documented abnormal cholesterol; abnormal fasting capillary glucose; abnormal angiogram; ECG or exercise stress tests or a diagnosis of diabetes mellitus; or any history suggestive of angina.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-10 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Vasomotor symptoms prospectively recorded in the final month of therapy by therapy assignment, with pre-therapy baseline vasomotor symptoms as a covariate. | Four months
Forearm blood flow by plethysmography prospectively measured before and after three months of therapy | Four months

SECONDARY OUTCOMES:
Other hormone-related quality of life measures on the Daily Menopause Diary®, especially self worth, sleep, and energy, recorded during the 4 months of the study. | Four months
Changes in two Quality of Life instruments - the Rand SF-36 and the Menopause-specific Quality of Life (MenQoL) questionnaires, measured at baseline and at the end of the study period | Four months
Lipid, blood pressure (BP), waist circumference and weight changes, measured at baseline and at the end of the study period | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Jerilynn Prior, Principal Investigator — University of British Columbia
Locations (1):
- Centre for Menstrual Cycle and Ovulation Research, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Prior JC, Elliott TG, Norman E, Stajic V, Hitchcock CL. Progesterone therapy, endothelial function and cardiovascular risk factors: a 3-month randomized, placebo-controlled trial in healthy early postmenopausal women. PLoS One. 2014 Jan 21;9(1):e84698. doi: 10.1371/journal.pone.0084698. eCollection 2014. PMID 24465425
- [Derived] Sathi P, Kalyan S, Hitchcock CL, Pudek M, Prior JC. Progesterone therapy increases free thyroxine levels--data from a randomized placebo-controlled 12-week hot flush trial. Clin Endocrinol (Oxf). 2013 Aug;79(2):282-7. doi: 10.1111/cen.12128. Epub 2013 May 6. PMID 23252963
- [Derived] Hitchcock CL, Prior JC. Oral micronized progesterone for vasomotor symptoms--a placebo-controlled randomized trial in healthy postmenopausal women. Menopause. 2012 Aug;19(8):886-93. doi: 10.1097/gme.0b013e318247f07a. PMID 22453200
- See also: Centre for Menstrual Cycle and Ovulation Research — http://www.cemcor.ubc.ca